CLINICAL TRIAL: NCT06285201
Title: A Phase 1 Clinical Study to Evaluate the Pharmacokinetic Comparability, Safety, Tolerability, and Immunogenicity of Felzartamab for Injection in Healthy Male Adult Subjects in China (Randomized, Double-blind, Crossover Design)
Brief Title: Study of Felzartamab in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: TJ202001BE104
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): T-R
  Interventions: Drug: T; Drug: R
- Group B (Experimental): R-T
  Interventions: Drug: T; Drug: R

INTERVENTIONS:
Drug: T — 8 mg/kg IV of Test drug manufactured by I-Mab Biopharma(Hangzhou)
Drug: R — 8 mg/kg IV of Test drug manufactured by Patheon Italia

SUMMARY:
A Phase 1 Clinical Study to Evaluate the Pharmacokinetic Comparability, Safety, Tolerability, and Immunogenicity of Felzartamab for Injection Pre- and Post-changes of Process in Healthy Male Adult Subjects in China (Randomized, Double-blind, Single-dose, Two-formulation, Two-sequence, Two-period Crossover Design)

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged ≥ 18 years and ≤ 50 years when signing the ICF.
* Weight ≥ 50 kg and ≤ 80 kg, with a BMI ≥ 19.0 and ≤ 28.0 kg/m2 (inclusive).
* The study doctor determines that the overall health status of the subject is good (normal or abnormal but not clinically significant) based on the subject's medical history, physical examinations, vital signs, ECG, and laboratory test results.
* Subjects who are voluntarily participate in the study, and can understand and sign the ICF.
* Subjects (including their partners) who have no plans for pregnancy or sperm donation during the study and within 6 months after the last dose, and voluntarily use effective contraceptive measures. Specific contraceptive measures are described in Appendix 4.

Exclusion Criteria:

* Subjects with diseases that may affect his safety or the results of the study, including but not limited to cardiovascular, respiratory, endocrine, metabolic, renal, hepatic, gastrointestinal, dermatological, infectious, malignant tumors, hematological, skeletal, genitourinary, neurological/psychiatric diseases, and are clinically significant in the opinion of the investigator.
* Subjects who have had acute, chronic, or potential infectious diseases within 1 month pre-dose.
* Subjects with known immune system diseases (such as autoimmune diseases or immunodeficiency diseases), including but not limited to autoimmune hemolytic anemia, etc.
* Subjects who have had a single episode of herpes zoster (shingles) involving the skin or central nervous system within the 6 months pre-dose.
* Subjects who currently have or have a history of multiple episodes of herpes zoster involving the skin or central nervous system.
* Subjects with chronic diarrhea or enteritis within 1 year pre-dose.
* Subjects with positive result for blood group antibody screening (IAT).
* Subjects who have received monoclonal antibodies, cell therapies within 6 months pre-dose, or have previously received daratumumab or similar drugs, or drugs targeting CD38.
* Subjects who have taken any medicine, including prescription drugs, over-the-counter drugs, and herbal medicine, within two weeks pre-dose.
* Subjects who are suspected or confirmed to be allergic to multiple drugs or foods, including drugs or drug excipients in this clinical study.
* Subjects who have a history of fear of needles or blood, or have difficulty with venous blood collection (have a history of difficulty with blood collection or have corresponding symptoms and signs, and cannot tolerate venous puncture).
* Subjects with the history of blood donation or blood loss of ≥ 200mL in total within 3 months pre-dose;
* Subjects who have participated in any other clinical studies of investigation drug or medical device within the 3 months pre-dose (or 5 half-lives for investigation drugs with so long half-life that the duration of its 5 half- lives is > 3 months).
* Subjects who have undergone major surgery within the last 3 months prior to signing the ICF.
* Subjects who are positive for Hepatitis B (positive for HBsAg or HBcAb and HBV-DNA levels of ≥ 500 cps/mL [or HBV-DNA ≥ 100 IU/mL]), HCV antibodies, HIV antibodies, and anti-TP antibodies.
* Smokers who have smoked more than 5 cigarettes per day in the 3 months prior to the study or who are unable to stop using any tobacco products during the study.
* Subjects who have received attenuated or live viral vaccines (such as Bacille Calmette-Guérin [BCG]) or viral vector vaccines within 12 months before the first dose of investigation drug, or plan to receive within 12 months post-dose.
* Subjects who have received vaccines other than attenuated or live virus vaccines, as well as virus vector vaccines talked above, such as inactivated vaccines, recombinant subunit vaccines, etc. within the 1 month before the first dose.
* The investigator determines the subjects have any other factors that make them unsuitable to participate in this study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Primary PK Endpoint | 36 days after dosing
  AUC0-∞

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojiao Li, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Jilin, Changchun, China

IPD SHARING:
Plan to Share IPD: No